CLINICAL TRIAL: NCT05731414
Title: Cognitive Behavioural Therapy Compared to Cognitive Remediation for Schizophrenia-Spectrum Disorders
Brief Title: Outcomes From Remediation and Behavioural Intervention Techniques
Acronym: ORBIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ontario Shores Centre for Mental Health Sciences (Other); Queen's University (Other); Centre for Addiction and Mental Health (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Best, Assistant Professor, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 43817
Record Dates: First submitted 2023-01-19; First posted 2023-02-16 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Psychosis; Psychotic Disorders; Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive a) individual CBT + group sham CR, b) group CR + individual Befriending, or c) individual CBT + group CR. Block, cohort randomization will be coordinated by the trial manager at the central site (UTSC), with stratification by treatment site. Cohorts of 5 participants will be randomized to one of the 3 treatment conditions in randomized block sizes of 4, 8, or 12 using a pre-specified randomization list.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This will be a double-blind (participant, assessor) trial. Participants will be informed that they will receive one individual session and one group session of treatment per week but will not be told which group they are assigned to. Participants will be instructed not to talk about their therapy to the assessor but if the assessor becomes aware of group allocation, then a new assessor will be assigned for all follow-up assessments. Due to the nature of the interventions, it is not possible for therapists to be blind to treatment condition, however, therapist fidelity to each intervention will be monitored through ratings on established fidelity measures. To protect against contamination separate therapists will deliver the active and control therapies.
  The Principal Investigator also remains blind to randomization, as the trial manager is the only one who has access to this.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Individual CBTp + Group Sham CR (Experimental): Individual formulation-based CBT will be delivered for one hour per week using a manual that has been validated in over 1000 individuals with schizophrenia-spectrum disorders across all stages of illness.
  Sham CR was developed by Dr. Best and Dr. Bowie (CI) to control for the non-specific effects of CR such as computer practice and group discussion.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Psychosis (CBTp); Behavioral: Sham Cognitive Remediation
- Group CR + Individual Befriending (Sham CBTp) (Experimental): Action-based cognitive remediation (ABCR) will be delivered in group sessions one hour per week. ABCR was developed by Dr. Bowie (CI) and Dr. Best (PI) and has been found efficacious for schizophrenia-spectrum disorders in three clinical trials.
  Befriending will be delivered according to a manual validated to control for the non-specific effects of CBT, such as duration of therapeutic contact, client expectancy effects, therapeutic alliance, and therapist warmth.
  Interventions: Behavioral: Cognitive Remediation Therapy (CR); Behavioral: Befriending
- Individual CBTp + Group CR (Experimental): Individual formulation-based CBT will be delivered for one hour per week using a manual that has been validated in over 1000 individuals with schizophrenia-spectrum disorders across all stages of illness.
  Action-based cognitive remediation (ABCR) will be delivered in group sessions one hour per week. ABCR was developed by Dr. Bowie (CI) and Dr. Best (PI) and has been found efficacious for schizophrenia-spectrum disorders in three clinical trials.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Psychosis (CBTp); Behavioral: Cognitive Remediation Therapy (CR)

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Psychosis (CBTp) — Individual formulation-based CBT will be delivered for one hour per week using a manual that has been validated in over 1000 individuals with schizophrenia-spectrum disorders across all stages of illness. This approach has demonstrated moderate to large improvements on symptoms and small to moderate effects on functioning. The first four sessions are devoted to building therapeutic rapport and developing collaborative treatment goals. The following phase focuses on developing formulations of why difficulties persist and using cognitive and behavioural change strategies. A longitudinal formulation is then offered to better understand how their difficulties developed. The final 2-4 sessions focus on consolidating the learning that occurred during treatment so that participants can maintain their improvement. Therapy homework is collaboratively assigned at the end of sessions to promote new learning in between sessions.
  Arms: Individual CBTp + Group CR; Individual CBTp + Group Sham CR
Behavioral: Cognitive Remediation Therapy (CR) — Action-based cognitive remediation (ABCR) will be delivered in group sessions one hour per week. ABCR was developed by Dr. Bowie (CI) and Dr. Best (PI) and has been found efficacious for schizophrenia-spectrum disorders in three clinical trials. ABCR involves practicing computerized training exercises with difficulty level dynamically titrated to improve neurocognitive abilities. Then participants engage in strategy discussions with other group members to develop new cognitive strategies. Finally, participants complete role-play simulations of real-world activities to practice their cognitive strategies in simulations of everyday life. ABCR is more effective for improving functioning than traditional approaches to CR. Homework consists of additional cognitive training and practicing cognitive strategies in everyday life.
  Arms: Group CR + Individual Befriending (Sham CBTp); Individual CBTp + Group CR
Behavioral: Befriending — Befriending will be delivered according to a manual validated to control for the non-specific effects of CBT, such as duration of therapeutic contact, client expectancy effects, therapeutic alliance, and therapist warmth. Befriending consists of 1-hour individual sessions once per week and involves a series of conversations similar to those one might have with a social acquaintance. These conversations involve discussion of neutral topics without problem-solving, coping strategies, or exploration of emotion. If emotional or mental health-related topics are brought up therapists redirect back to a neutral topic.
  Arms: Group CR + Individual Befriending (Sham CBTp)
Behavioral: Sham Cognitive Remediation — Sham CR was developed by Dr. Best and Dr. Bowie (CI) to control for the non-specific effects of CR such as computer practice and group discussion. Participants practice similar computerized exercises to ABCR, however, the exercises do not increase in difficulty. Participants then discuss enjoyment of the exercises but any discussion of cognitive strategies is redirected back to a neutral topic. We have previously found this condition to be an effective control for CR, with similar engagement to the active training group.
  Arms: Individual CBTp + Group Sham CR

SUMMARY:
It is currently unknown what factors predict response to Cognitive Behavioural Therapy for Psychosis (CBTp) or Cognitive Remediation Therapy (CR) among individuals with schizophrenia-spectrum disorders, thus the current trial will examine predictors of response to determine who requires the combined intervention and who might respond sufficiently to either monotherapy.

DETAILED DESCRIPTION:
Dominant treatment approaches for schizophrenia-spectrum disorders improve psychiatric symptoms but do little to improve community functioning, leading to persistent disability and substantial economic burden. The proposed trial aims to examine the efficacy of a multi-mechanism approach to combining CBT and CR with the goal of predicting treatment response to either monotherapy or combination therapy. To date, there have been no randomized controlled trials examining the combination of CBT and CR. Given the differential mechanisms of CBT and CR, the combined multi-mechanism approach is expected to more effectively improve functional recovery than either monotherapy. Additionally, it is currently unknown what factors predict response to CBT or CR, thus the current trial will examine predictors of response to determine who requires the combined intervention and who might respond sufficiently to either monotherapy. The proposed trial will be one of the largest trials of psychosocial interventions for schizophrenia-spectrum disorders ever conducted and will simultaneously evaluate the combined intervention and moderators of differential treatment response. Narrower fields of inquiry examining mono-mechanism interventions have demonstrated little utility in improving functional recovery in schizophrenia, thus, the proposed approach represents a critical advancement by examining the utility of a multi-mechanism cognitive intervention and determining characteristics of those requiring this level of treatment.

The goals of the current study are three-fold:

1. Examine the efficacy of combining CBT and CR on the primary outcome of community functioning, and secondary outcomes of quality of life, personal recovery, psychiatric symptoms, and neurocognition compared to either intervention alone.
2. Examine demographic, cognitive, and psychological factors that predict differential response to CBT, CR, or combined CBT and CR.
3. Examine the specificity of cognitive content and cognitive functions as therapeutic mechanisms in CBT and CR respectively.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Diagnosed with schizophrenia-spectrum disorders
* Can read, write, and speak English

Exclusion Criteria:

* Neurodevelopmental disability or neurocognitive disorder
* CBT or CR in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Social Functioning Scale (SFS) | Change between baseline assessment and 18-month assessment
  The Social Functioning Scale (SFS) is an interview-based measure assessing basic social adjustment skills. It can be administered to both the participant and informants. Seven aspects are evaluated: (1) social engagement/withdrawal (with raw scores ranging from 0-15); (2) interpersonal behavior (with raw scores ranging from 0-9); (3) pro-social activities (with scores ranging from 0-66); (4) recreation (with scores ranging from 0-45); (5) independence-competence (with scores ranging from 0-39); (6) independence-performance (scores ranging from 0-39); and (7) employment/occupation (with scores ranging from 0-10). The lowest total score would be a 0 while the highest would be a 223. Higher scores are indicative of better social functioning.

SECONDARY OUTCOMES:
World Health Organization Quality of Life Scale Brief Version (WHOQOL-BREF) | Change between baseline assessment and 18-month assessment
  The WHOQOL-BREF is a 26-item self-report measure assessing quality of life. The four domains included are: (1) physical health, (2) psychological, (3) social relationships and (4) environment. Responses are rated on a 5-point scale, and reverse-scored items are included. The highest total raw score would be a 130, while the lowest would be a 26. Higher scores indicate better quality of life.
Questionnaire About the Process of Recovery (QPR) | Change between baseline assessment and 18-month assessment
  QPR is a self-report measure assessing recovery with people experiencing psychosis. This version contains 22 items while the response to each statement is scored on a 5-point Likert scale ranging from "0 = strongly disagree" to "4 = strongly agree". The lowest possible score is 0 and the highest score could be 88. Higher scores would indicate better recovery.
Positive and Negative Syndrome Scale (PANSS) | Change between baseline assessment and 18-month assessment
  The PANSS is a 30-item semi-structured interview assessing positive, negative symptoms and general psychopathology. Each item is scored on a 7-point scale (1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderate severe, 6 = severe, 7 = extreme). The lowest score would be a 30 and the highest score would be 210. A higher score would indicate increased symptomology. A 15-point change on the PANSS is associated with clinically meaningful change.
Psychotic Symptom Rating Scale (PSYRATS) | Change between baseline assessment and 18-month assessment
  The PSYRATS assesses frequency and distress associated with the experiences of auditory hallucinations and delusions based on the PANSS interview. Each of the 17 items is scored on a 5-point scale, where a score of 0 indicates no presence, and 4 indicates the highest severity. The lowest score would be a 0 and the highest score would be 68. A higher score would indicate increased symptomology.
Neurocognitive Assessment | Change between baseline assessment and 18-month assessment
  Neurocognition will be assessed using a cognitive batter that assess the MATRICS cognitive domains. Assessments include Oral Trail Making Test, Hopkins Verbal Learning Test, Letter Number Span, WMS Symbol Span, Brief Visuospatial Memory Test, DKEFS Verbal Fluency, Hinting Task, CNS Vital Signs Symbol Digit Coding, CNS Nonverbal Reasoning, CNS 4-part CPT. A Neurocognitive Composite score will be calculated based on these subtests. Z-scores will range between -3.00 and +3.00, with higher scores indicating better performance.
Beliefs About Paranoia Scale (BAPS) | Change between baseline assessment and 18-month assessment
  The BAPS is a 31-item self-report measure assessing metacognitive beliefs about paranoia. The degree of agreement to each statement is scored on a 4-point scale (1 = not at all, 2 = somewhat, 3 = moderately so, 4 = very much). Scales include positive, negative and normalizing beliefs about paranoia, and paranoia as a survival strategy. The lowest score would be 31 and the highest score would be 124. Higher scores are indicative of more beliefs and are shown to be related to paranoid ideation.
Interpretations of Voices Inventory (IVI) | Change between baseline assessment and 18-month assessment
  The IVI is a 26-item self-report measure assessing perceptions of auditory hallucinations. Meta-physical beliefs about voices, positive beliefs about voices, and beliefs about loss of control are evaluated. Responses are rated on a 4-point scale (1 = Not at all, 2 = Somewhat, 3 = Moderately so, 4 = Very much). The lowest score would be a 26 while the highest score would be a 104. Higher scores are indicative of more and stronger beliefs.
Brief Core Schema Scale (BCSS) | Change between baseline assessment and 18-month assessment
  The BCSS is a 24-item self-report measure assessing positive and negative judgments individuals hold about themselves and others. Responses are first given dichotomously as "no" or "yes". "No" is scored as 0 and if the answers are "yes", the intensity of beliefs are then rated on a 4-point scale (1 = believe it slightly, 2 = believe it moderately, 3 = believe it very much, 4 = believe it totally). The lowest score would be a 0 and the highest score would be a 96. Higher scores in the positive-self subscale indicate more positive beliefs about selves, while higher scores in the negative-self subscale indicate more negative beliefs about selves. Higher scores in the positive-others subscale indicate more positive beliefs about others, while higher scores in the negative-others subscale indicate more negative beliefs about others.
Defeatist Beliefs Scale (from Dysfunctional Attitudes Scale, DAS) | Change between baseline assessment and 18-month assessment
  The rating format for the 80 Dysfunctional Attitudes Scale items is a 7-point Likert scale ranging from totally agree to totally disagree. Possible responses are scored from 1 to 7, with the direction depending on whether agreement or disagreement with a particular belief is judged to be a maladaptive response, and with higher scores indicating more distorted thinking.
Treatment Inventory of Costs in Patients in Psychiatric Disorders (TiC-P) | Change between baseline assessment and 18-month assessment
  The TiC-P measures direct and indirect costs of health conditions.
  The first part contains 21 questions assessing healthcare costs, calculated by multiplying numbers of access with prices.
  The second part contains 12 questions assessing productivity losses. For paid work, productivity losses due to absence are measured by cost prices, with the number of workdays multiplying hours per day and a standard hourly rate. Scores on short-term absence are adjusted with long-term absence to avoid double-counting, while the friction period and measurement times are considered for scores on long-term absence. Productivity losses due to presenteeism are calculated by multiplying the number of workdays impaired with (1 - efficiency score/10) and hours per workday. Unpaid productivity losses are calculated by multiplying the days missed by the number of hours per day needed to make up the work, and a standard hourly rate.
  Higher scores indicate higher costs related to health conditions.
Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS) | Change between baseline assessment and 18-month assessment
  The SSTICS is a 21-item self-report measure assessing subjective cognitive complaints among patients with Schizophrenia. Frequency of experiencing each item is rated on a 5-point scale, ranging from "0 = Never" to "4 = Very Often". The lowest score would be a 0 and the highest score would be an 84. Higher scores are indicative of more subjective cognitive difficulties.
Davos Assessment of Cognitive Biases in Schizophrenia (DACOBS) | Change between baseline assessment and 18 month assessment
  DACOBS is a 42-item self-report inventory assessing cognitive processing biases associated with psychosis. The degree of agreement to each statement is scored on a 7-point Likert scale, ranging from "1 = strongly disagree" to "7 = strongly agree". The lowest score would be a 42 and the highest score would be a 294. Higher scores would indicate more cognitive biases.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Best, PhD, C.Psych, Principal Investigator — University of Toronto Scarborough
Locations (2):
- Canada (2):
  - University of Toronto Scarborough, Scarborough Village, Ontario
  - Ontario Shores Centre for Mental Health Sciences (Ontario Shores), Whitby, Ontario

IPD SHARING:
Plan to Share IPD: No